CLINICAL TRIAL: NCT04977505
Title: Absorption Rate and Bone Ingrowth of Absorbable Anchors Used in Shoulder Dislocation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021132
Record Dates: First submitted 2021-06-27; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-06

CONDITIONS: Shoulder Dislocation
Keywords: anterior dislocation; anchor
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pushlock: Patients with recurrent shoulder dislocation received surgery fixed by pushlock
  Interventions: Device: pushlock
- Gryphon: Patients with recurrent shoulder dislocation received surgery fixed by Gryphon
  Interventions: Device: gryphon

INTERVENTIONS:
Device: pushlock — The surgery procedure was performed with pushlock for fixation
  Groups: Pushlock
Device: gryphon — The surgery procedure was performed with Gryphon for fixation
  Groups: Gryphon

SUMMARY:
This study aims to analyze the absorption rate of Pushlock anchors and Gryphon anchors and the bone ingrowth of the anchor channel by consulting the postoperative CT images of patients with recurrent shoulder dislocation completed by myself. The investigators will analyze the influence factors of anchor absorption and bone ingrowth, which will provide a reference for improving anchor design and the improvement of surgical techniques.

DETAILED DESCRIPTION:
"Recurrent anterior dislocation of the shoulder joint is a common disease of the shoulder joint. The standard treatment methods include soft tissue repair surgery and bone tissue repair surgery. The former refers to arthroscopic labral suture (Bankart repair surgery), and the latter includes Latarjet surgery, Bristow surgery and Cuistow surgery pioneered by our team. Whether it is soft tissue repair surgery or bone tissue repair surgery, anchors are required for suture fixation during the operation.

The anchors currently in use include non-absorbable anchors and absorbable anchors. Non-absorbable anchors include metal anchors and peek material anchors, which remain in the body forever after the operation and cannot be absorbed. The absorbable anchors, in theory, will be absorbed 2 years after surgery.

Non-absorbable anchors have inherent limitations that limit their use. If the non-absorbable anchor loosens and shifts, it can cause severe cartilage damage. If complications such as re-dislocation occurred, revision surgery is required. Revision surgery is complicated because the non-absorbable anchor inserted in the initial surgery occupies the best anchor position. Metal anchors can cause artifacts and affect postoperative MRI imaging.

Therefore, absorbable anchors have gradually become routinely used in shoulder joint dislocation surgery.

The anchors currently used in our hospital for shoulder joint instability include Pushlock anchors from Arthrex and Gryphon anchors from Depuy Mitek. The materials are PLLA/β-TCP and PLGA/β-TCP. The absorption anchor starts to absorb in 1 year and completes absorption in about two years. The anchor tunnel will be filled with bone tissue. However, the investigators have found that the anchor cannot be wholly absorbed as scheduled. During the revision surgery, the original absorbable anchor can still be seen. Clear anchor tunnels can also be seen in CT films after 2 years postoperatively.

Published literature also show that the degradation rate of absorbable anchors is not the same. The literature report that anchors have not completed degradation and bone ingrowth within the time advertised by the manufacturers.

In summary, this study aims to analyze the absorption rate of Pushlock anchors and Gryphon anchors and the bone ingrowth of the anchor tunnel by consulting the postoperative CT films of subjects with recurrent shoulder dislocation completed by myself. The factors that affect anchor absorption and bone ingrowth provide a reference for improving anchor design and the improvement of surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* (1) The subject underwent Cuistow surgery, Bristow surgery, Latarjet surgery or Bankart surgery.
* (2) The surgeon was chief physician Cui Guoqing.
* (3) Pushlock anchor (2.9mm) or Gryphon anchor (3.0mm) was used during the operation, and the placement position was the glenoid.

Exclusion Criteria:

* (1) Ipsilateral shoulder joint, with a history of surgery.
* (2) Subjects with postoperative infection.
* (3) Subjects with incomplete data (no immediate postoperative CT or no postoperative CT films for more than 2 years).
* (4)Subjects with diabetes.
* (5)Revision surgery for shoulder dislocation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent Cuistow surgery, Bristow surgery, Latarjet surgery or Bankart surgery in Peking University Third Hospital for fixing the dislocated shoulder.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
hounsfield unit of anchor tunnel | 2 years after surgery
  It is an index used to evaluate the status of bone resorption. It was recorded of last CT films.
the diameter of anchor tunnel | 2 years after surgery
  It is an index used to evaluate the status of bone resorption. It can be measured in the last CT films.
Hounsfield unit of ossification site | 2 years after surgery
  It is an index used to evaluate the status of bone resorption. It was recorded of last CT films.

SECONDARY OUTCOMES:
unossified area of anchor tunnel | 2 years after surgery
  It is an index used to evaluate the status of bone resorption. It can be measured in the last CT films.
ossification quality score | 2 years after surgery
  It is a standard score used to qualify the status of ossification.

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No